CLINICAL TRIAL: NCT05220709
Title: Bio Impedance Monitoring as a Tool to Assess Fluid Status in the Pediatric Surgical Patient: Can we Measure a Fluid Shift
Brief Title: Bio Impedance Monitoring as a Tool to Assess Fluid Status in the Pediatric Surgical Patient? (PedFluid Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Vera Saldien, Principal Investigator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0576; 002090 (Other: Edge)
Record Dates: First submitted 2021-12-06; First posted 2022-02-02 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Fluid and Electrolyte Imbalance; Body Weight Changes; Children, Only
Keywords: bio impedance spectroscopy
MeSH Terms: conditions — Body Weight Changes

STUDY DESIGN:
Intervention Model Description: This is a single-centre pilot study to evaluate the feasibility of bio impedance measurements to determine fluid shifts in the pediatric population after a surgical procedure was performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bio impedance spectroscopy in children scheduled for elective surgery under general anesthesia (Other): All subjects receive bio impedance monitor measurements pre operatively and post operatively.
  Interventions: Diagnostic Test: bio impedance spectroscopy by means of the Body Composition Monitor (Name of the device is BCM from Fresenius Medical Care D GmbH)

INTERVENTIONS:
Diagnostic Test: bio impedance spectroscopy by means of the Body Composition Monitor (Name of the device is BCM from Fresenius Medical Care D GmbH) — The Body Composition Monitor provides information about the hydration status by a bioimpedance spectroscopy measurement of the body composition from which the level of overhydration can be derived. Four electrodes are used per measurement. All subjects get electrodes attached, following the wrist-ankle approach, in a tetrapolar arrangement. Two electrodes are placed on the hand: one on the wrist, and the second on the dorsal side of the metacarpalia, close to the phalanges. The other two electrodes are placed on the foot: one on the ankle, and the second on the dorsal side of the metatarsals, close to the phalanges of the toes. Age, gender, height, weight and blood pressure are registered in the device before starting the measurement. If the quality calculated by BCM is < 60%, the measurement will be repeated again. Measurements are taken under supervision of a trained technician or nurse.

SUMMARY:
The baseline infusion rate during surgery for pediatric patients still is the 'Holliday and Segar' rule (also known as the 4/2/1 rule) The question arises if this rule is not outdated, since it was calculated based on the caloric need of the pediatric population, calculated for cow milk. The study tends to validate the use of bio impedance measurements for registering fluid shifts in the pediatric surgical patients.

DETAILED DESCRIPTION:
The Body Composition Monitor (BCM, Fresenius Medical Care, Germany) is the first device that determines individual fluid status and body composition in an easy and objective way. The technology uses bioimpedance spectroscopy (BIS) to determine total body water (TBW) and extracellular water volume (ECW).It measures at 50 frequencies over a range from 5 to 1000 kHz to determine the electrical resistances of the total body water and the extracellular water. While high-frequency current passes through the total body water, low-frequency current cannot penetrate cell membranes and thus flows exclusively through the extracellular water.

To obtain the clinically relevant output parameters, two advanced physiological models are used in the BCM: a volume model, describing electrical conductance in a cell suspension enabling the total body water and extracellular water as well as the intracellular water (ICW) to be calculated, and a body composition model calculating the three principal body compartments overhydration, lean tissue and adipose tissue from ECW and TBW information.

The measurement is a non-invasive and accurate method that is easy to apply and results are obtained within just two minutes. It has been extensively used in patients with kidney disease receiving dialysis, both in adult and pediatric patients. However, bio impedance spectrometry has not yet been tested in the perioperative setting.

This is a single-center pilot study to evaluate if bio impedance measurement is a workable tool to determine fluid shifts in the pediatric population after a surgical procedure was performed under general anesthesia. Patients will be seen preoperatively by an anesthesiologist which is standard of care upon surgery under general anesthesia and eligibility will be evaluated. Informed consent will be asked and has to be signed by the accompanying parent or legal guardian. Where possible, care will be taken to inform the child itself about the content of the study and to get a written acknowledge. There are no other investigations necessary for this research. All patients on the day of surgery will be fasted as by the guidelines of the European Society of Anesthesia. For patients in daycare surgery, measurements with BCM will be performed preoperatively and postoperatively before ending the IV line on the ward. For inpatient hospitalisation, measurements by BCM will be performed preoperatively, postoperatively 6 hours after induction and postoperatively 24 h after induction.. Age, gender, height, weight and blood pressure are registered in the device before starting the measurement. If the quality calculated by BCM is < 60%, the measurement will be repeated again and only good quality measurements will be used.

Data are collected on chip cards by the BCM. Data can be transferred to a personal computer for further analysis with the Fluid Management Tool (FMT). Site requirements is the availability of a low electronic surrounding for correct measurement. After discharge of the hospital no further follow up assessments regarding this study are needed.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery or investigation under general anesthesia
* Day care or inpatient hospitalisation

Exclusion Criteria:

* If sedation is needed instead of general anesthesia
* Critically ill patients for urgent surgery
* Patients who cannot lie still for performing correct measurements on the bio impedance monitor
* No informed consent obtained

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
total body water | measurements with BCM will be done pre-surgery
  sum of intracellular water and extracellular water, calculated in liter
total body water | measurements with BCM will be done within 6 hours post-surgery for patients in day care
  sum of intracellular water and extracellular water, calculated in liter
total body water | measurements with BCM will be done within 24 hours post-surgery for hospitalized patients
  sum of intracellular water and extracellular water, calculated in liter

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD,PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium